CLINICAL TRIAL: NCT05605639
Title: Phrenic Afferences In Organic and Metabolic Illness: Central Sensitization
Brief Title: Phrenic Nerve Infiltration in Neck Pain
Acronym: PAINOMICS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Angel Oliva Pascual-Vaca, Dr., University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0746-N-21
Record Dates: First submitted 2022-10-23; First posted 2022-11-04 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Chronic Neck Pain
Keywords: phrenic nerve; anesthesia, local
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phrenic nerve anesthetics infiltration (Experimental): The experimental intervention will consist of ultrasound-guided anesthetic blockade of the phrenic nerve at the laterocervical supraclavicular level with 1 ml of lidocaine without vasoconstrictor 2% to infiltrate the skin and 3ml of bupivacaine without vasoconstrictor 0.25% for neural blockade, making the local anesthetic surround the nerve between the anterior scalene muscle and the sternocleidomastoid muscle.
  Interventions: Drug: Bupivacaine
- Physiological serum infiltration (Placebo Comparator): The placebo intervention will be similar in relation to 2% lidocaine without vasoconstrictor for the skin, but an ultrasound-guided puncture will be performed at the level of the subcutaneous cellular tissue by injecting 3 ml of physiological saline.
  Interventions: Other: Placebo (physiological saline serum infiltration)

INTERVENTIONS:
Drug: Bupivacaine — The experimental intervention will consist of ultrasound-guided anesthetic blockade of the phrenic nerve at the laterocervical supraclavicular level with 1 ml of lidocaine without vasoconstrictor 2% to infiltrate the skin and 3ml of bupivacaine without vasoconstrictor 0.25% for neural blockade, making the local anesthetic surround the nerve between the anterior scalene muscle and the sternocleidomastoid muscle.
  Other Names: Bupivacaine B. Braun 2.5 mg/ml
  Arms: Phrenic nerve anesthetics infiltration
Other: Placebo (physiological saline serum infiltration) — The placebo intervention will be similar in relation to 2% lidocaine without vasoconstrictor for the skin, but an ultrasound-guided puncture will be performed at the level of the subcutaneous cellular tissue by injecting 3 ml of physiological saline.
  Arms: Physiological serum infiltration

SUMMARY:
Neck pain frequently present comorbidities in peridiaphragmatic organs. The innervation of these organs include the phrenic nerve. It is known that peridiaphragmatic organs trigger referred pain in the neck area. As well, previous studies have shown that visceral disorders increase sensitization in somatic tissues. This study aims to analyze the ability of phrenic nerve infiltration to diminish sensitization and improve neck symptoms in the absence of neurological, traumatic or infectious pathology that justifies the pain, by means of a randomized controlled trial.

DETAILED DESCRIPTION:
Pain is a major problem due to issues such as the impact on quality of life and the associated health and social costs. Neck pain is a very common disorder in our society. It is characterized by the presence of hyperalgesia, increased muscle tone, limited range of motion and sensitization. It is well known that pain of visceral origin can generate all these phenomena. In most cases, there is no antecedent of trauma, and no evidence of a specific origin (oncologic, rheumatic, infectious…), so patients are classified as suffering non-specific or idiopathic pain. The absence of a specific diagnosis makes it difficult to find a therapeutic target to increase the probability of successful therapies. Thus, in the case of neck pain, the recurrence of consultations is very high.

It is known that cervical pain frequently presents peridiaphragmatic visceral comorbidities. Furthermore, it is known that these peridiaphragmatic organs produce referred pain to the neck, and this pain is known as phrenic pain. To date, there are no studies that analyze the role of phrenic afferents in subjects with neck pain and peridiaphragmatic visceral disorders. The aim of this study is to evaluate the effect of phrenic nerve anaesthesia in subjects with neck pain. For this purpose, the investigators intend to perform a randomised clinical trial, assessing the effects on pain threshold to pressure, visual analogue scale, range of motion and craniocervical questionnaires. There will be only one intervention session. The experimental group will receive an ultrasound-guided anaesthetic infiltration of the phrenic nerve, while the control group will receive a placebo infiltration. A one-week follow-up, with intermediate measurements, will be carried out to assess the evolution of cervical sensitization and symptomatology.

The results of this study will make it possible to establish the role of peridiaphragmatic organic disorders and phrenic afferents in cervical pain, thus making it possible to specify a specific therapeutic target (phrenic nerve) as well as the importance of visceral treatment in subjects presenting for consultation for cervical pain.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 and under 64 years old
* Patients attending to the physician or physical therapist with a main complaint of neck pain
* Presentation of any peridiaphragmatic visceral disorder.
* That the subject agrees to participate in the project by signing the informed consent.

Exclusion Criteria:

* Illness of neurological, traumatic, oncological, infectious or rheumatic (fibromyalgia, ankylosing spondylitis...) origin.
* Uncooperative subject.
* Severe psychiatric illness.
* Loss of Cognitive Ability.
* Contraindication to infiltration of the phrenic nerve.
* History of head, spinal or upper limb surgery
* History of infiltration for the neck pain in the previous 3 months
* History of physical therapy for the neck pain in the previous 30 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in algometry | Pre-intervention. Post-intervention: 1 hour, 2 hours, 3 days and 7 days
  Pressure pain threshold in neck tissues. PPT levels defined as the minimum necessary pressure to evoke pain will be evaluated using a handheld electronic pressure algometer.

SECONDARY OUTCOMES:
Range of motion | Pre-intervention. Post-intervention: 1 hour, 2 hours, 3 days and 7 days
  Neck range of motion.The range of motion will be assessed in degrees. Flexion, extension, left and right side flexion, and left and right rotation will be assessed, and the sum of all of those parameters will be the considered outcome.
Visual Analogue Scale | Pre-intervention. Post-intervention: 1 hour, 2 hours, 3 hours, 6 hours, 24 hours, 2 days, 3 days and 7 days
  Perceived neck pain. Self-perceived pain intensity will be evaluated during all active cervical movements by a 0 to 10 Visual Analogue Scale (VAS), where 0 denotes no pain and 10 denotes the maximum possible pain.
Neck Disability Index | Pre-intervention. Post-Intervention: 3 days and 7 days.
  Neck Disability Index (Questionnaire). The Neck Disability Index will be used in the Spanish version. This questionnaire assesses how neck pain affects the ability to manage everyday-life activities. Scores range from 0-50 with higher scores indicating higher disability.
Headache Impact Test-6 | Pre-intervention. Post-intervention: 3 days and 7 days.
  Headache Impact Test (Questionnaire). The Headache Impact Test-6 was developed to measure a wide spectrum of the factors contributing to the burden of headache, and it has demonstrated utility for generating quantitative and pertinent information on the impact of headache. Scores range from 0-120 with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Oliva Pascual-Vaca, Dr, Principal Investigator — University of Seville
Locations (2):
- Spain (2):
  - Nacho Navarro Fisioterapia, Dos Hermanas, Seville
  - Crux Roxa, Seville

IPD SHARING:
Plan to Share IPD: No